CLINICAL TRIAL: NCT03526705
Title: The Effect of NB-UVB on Interleukin-36 Levels in Psoriasis Lesional Skin
Brief Title: The Effect of NB-UVB on Interleukin-36 Levels in Psoriasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina Saadi, Lecturer, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Kapu1
Record Dates: First submitted 2018-05-04; First posted 2018-05-16 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nb-uvb (Experimental): psoriasis patients will receive 26 sessions of nb-uvb phototherapy
  Interventions: Device: NB-UVB

INTERVENTIONS:
Device: NB-UVB — Phototherapy

SUMMARY:
Psoriasis is an immune-mediated skin disease that affects 1-2 % of the population. Several cytokines have been found to be involved in the complex pathogenesis of this disease. Il- 36 is one of the cytokines sharing in psoriasis pathogenesis, as its levels are elevated in psoriatic plaques. Cathepsin G is known to activate Il- 36 and promote inflammation in psoriasis.NB-UVB is one of the important treatment modalities for psoriasis.

The aim of this study is to detect the effect of NB-UVB on the lesional levels of IL-36 in psoriasis.

DETAILED DESCRIPTION:
25 psoriasis patients will receive 26 sessions of phototherapy (NB-UVB). Patients will receive 3 sessions per week. Tissue levels of IL-36 and Cathepsin G will be assessed in skin lesions before starting treatment and after completing the 26 sessions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with psoriasis vulgaris of both sexes
* Age between 18 and 60 years old.

Exclusion Criteria:

* Pregnant females
* Patients receiving systemic treatment or topical treatment for psoriasis within the past two months.
* Patients having other dermatological diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-07-15 (Estimated); Primary Completion 2020-01-15 (Estimated); Study Completion 2020-01-15 (Estimated)

PRIMARY OUTCOMES:
changes in Il-36 levels in 25 psoriasis patients after 26 sessions of NB-UVB | 6 months
  primary

SECONDARY OUTCOMES:
changes in cathepsin G levels in 25 psoriasis patients after 26 sessions of NB-UVB psoriasis | 6 months
  secondary

IPD SHARING:
Plan to Share IPD: No